CLINICAL TRIAL: NCT03803501
Title: Effectiveness of a Condensed Functional Restoration Program for Patients With Chronic Low Back Pain: a Study of 193 Patients
Acronym: PRAMH
Status: Completed | Type: Observational
Sponsor: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, Thomas Davergne, Physiotherapist, Master of Science and PhD candidate, principal investigator, Pitié-Salpêtrière Hospital
Other Study IDs: HSalpetrierePRAMH
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: condensed functional restoration program — The condensed functional restoration program (CFRP) is a complex multidisciplinary intervention proposed as usual care according to international guidelines. The program takes place in our department of rheumatology, 6 hours per day, 1 day a week, for 4 weeks. Patients are included during consultation or Hospitalisation and are in groups of 6 maximum per FRP. The CRFP was developed on the basis of therapeutic patient education programs and physical exercises (Van Wambeke 2017, Desthieux 2014). Three hours per day are devoted to physical exercises which were divided into three periods: warming, stretching, and muscular strengthening. Specific exercises adapted to work circumstances (like manutention) are taught. Muscular strengthening is based on isotonic contraction on fitness devices. Education is based on 1 hour long educative session adapted from back school programs once a week. Educative booklets are also given to the patients.
  Other Names: multidisciplinary rehabilitation program

SUMMARY:
The aim was to assess the effectiveness of a condensed functional restoration program (CFRP) for patients with chronic low back pain and professional activity.

Methods: Longitudinal 1 to 3 months study of patients with non-specific chronic low back pain in one tertiary care hospital, participating in a CFRP (complex interprofessional intervention over 4 days). The primary outcome was the Oswestry Disability Index (ODI) (0-100 scale). Secondary outcomes included pain, quality of life (EQ5D), patient acceptable symptom state, presenteeism, absenteeism and psychological distress (Hospital Anxiety and Depression scale). Outcomes were compared using paired sample Student's t-test or Chi2 between baseline and last follow-up. Logistic regression was used to identify factors associated with better response (improvement of ODI higher than 12.8) and included baseline demographic, psychological and physical assessment variables.

ELIGIBILITY:
Inclusion Criteria:

* non-specific cLBP (>3 months) with or without radicular pain, not currently in prolonged sick leave, no current indication for surgery, fluent in French, difficulties to maintain daily physical activity due to LBP with Oswestry Disability Index and lumbar and radicular pain at baseline and at end of intervention or 3-month follow-up available.

Exclusion Criteria:

* specific LBP and organic contraindication to physical exercise.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with chronic low back pain who participated in the condensed functional restoration program between April 2012 and April 2018
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  gives a subjective percentage score of level of function (disability) on a 0 to 100 scale, 100 being the highest disability state

SECONDARY OUTCOMES:
lumbar pain | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  visual analogue scale (0-100)
Radicular pain | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  visual analogue scale (0-100)
quality of life | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  EQ5D scale, converted into a global index score with 1 indicating no restriction of quality of life and -1 the worse quality of life possible
patient acceptable symptom state | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  where patients reported their satisfaction on state of symptoms by picking "acceptable" or "non acceptable"
World Health Organisation Health and Work Performance Questionnaire for absolute presenteeism | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  (reflecting the patient's overall job performance on the days worked during the past 4 weeks, 0-100, 100 being the highest amount of performance)
relative absenteeism | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  (rapport between the hours lost and the hours expected to work per month, 0-100, 100 indicates the higher amount of absenteeism)
psychological distress | change between baseline score and last follow-up data, i.e. data at 3 months follow-up or score at end of intervention if not available
  (Hospital Anxiety and Depression scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Davergne Thomas, Paris, France

IPD SHARING:
Plan to Share IPD: No